CLINICAL TRIAL: NCT04569864
Title: Comparing Mild Versus Moderate Hypothermic Circulatory Arrest With Unilateral Anterograde Cerebral Perfusion in Hemiarch Replacement
Brief Title: Mild vs Moderate Hypothermic Circulatory Arrest With Unilateral Anterograde Cerebral Perfusion in Hemiarch Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Erdeni L. Sonduev, Study Investigator and Coordinator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hypothermia
Record Dates: First submitted 2020-09-19; First posted 2020-09-30 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Intervention Model Description: The total patient population will be randomized into 2 groups. The first group of the patients during aortic hemiarch replacement, mild hypothermia (30-32°C) will be used during circulatory arrest. (main group). The second group of the patients during aortic hemiarch replacement, moderate hypothermia (26-28°C) will be used during circulatory arrest. (control group).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild hypothermia (30-32°C) (Experimental): During aortic hemiarch replacement, mild hypothermia (30-32°C) will be used during circulatory arrest.
  Interventions: Procedure: Hypothermic circulatory arrest with unilateral selective anterograde cerebral perfusion
- Moderate hypothermia (26-28°C) (Active Comparator): During aortic hemiarch replacement, moderate hypothermia (26-28°C) will be used during circulatory arrest.
  Interventions: Procedure: Hypothermic circulatory arrest with unilateral selective anterograde cerebral perfusion

INTERVENTIONS:
Procedure: Hypothermic circulatory arrest with unilateral selective anterograde cerebral perfusion — Hypothermic circulatory arrest provides protection to cerebral and visceral organs.

SUMMARY:
The aim of our study is to analyze the immediate and long-term results between patients undergoing hemiarch replacement with ACP under mild hypothermic (30-32 °C) circulatory arrest versus moderate hypothermic (26-28 °C) circulatory arrest. It is hypothesized that circulatory arrest using mild hypothermia (30-32°C) and uSACP will result in complications reduction, during aortic hemiarch replacement, when compared to moderate hypothermia (26-28°C) and uSACP. For this purpose all of the patient population will be randomized into 2 groups. The first group of the patients during aortic hemiarch replacement, mild hypothermia (30-32°C) will be used during circulatory arrest. The second group of the patients during aortic hemiarch replacement, moderate hypothermia (26-28°C) will be used during circulatory arrest.

DETAILED DESCRIPTION:
Mild versus moderate hypothermic circulatory arrest during aortic hemiarch replacement Hypothermic circulatory arrest with unilateral selective anterograde cerebral perfusion (SACP) is an important surgical technique, allowing complex aortic surgeries to be performed safely. One of the main positive aspects of the strategy for changing the hypothermia temperature is to reduce the systemic inflammatory response, minimize visceral organ dysfunction, and reduce the risk of postoperative bleeding - the adverse effects of hypothermia Patients will be operated for ascending aortic aneurysm in a hypothermic circulatory arrest with unilateral SACP. The main difference is during aortic hemiarch replacement, moderate hypothermia (26-28°C) and mild hypothermia (30-32°C) will be used during circulatory arrest. All data will be prospectively collected and recorded. All surgeries will be perform concurrently in the same time period. Experienced in aortic pathology surgeons will perform these operations.

Description of the procedures:

All surgical procedures will be performed via median sternotomy. During the aortic arch anastomosis, continuous, unilateral SACP using innominate artery will be employed. Unilateral SACP may be converted to bilateral ACP at the surgeon's discretion if adequate cerebral flows are not achieved or if there are concerns with cerebral oximetry measurements.

Once on CPB, the patient will be cooled to a nasopharyngeal (NP) temperature of either 30-32 °C or 26-28 °C, depending on to which treatment arm the patient has been randomized. Rectal temperature with be monitored as an additional temperature sites. Unilateral SACP will only be initiated once the target temperature has been reached. SACP via the innominate artery will be commenced with target flows of 8-10 ml/kg/min and perfusion pressure of 60-80 mmHg. Perfusion adequacy will be evaluated using measurement of blood pressure in both radial arteries and cerebral oximetry using near-infrared spectroscopy (NIRS).

After completion of the aortic hemiarch replacement, CPB will be resumed and the patient re-warmed to 36 °C prior to coming off CPB, with a = 1 °C temperature difference between temperature monitoring sites (NP and rectal).

Intraoperative information will be collected from the anesthetic record, surgical notes and perfusion records. Intraoperative data collection will include total operative time, CPB time, cross-clamp time, hypothermic cardiac arrest time, uSACP time, lowest nasopharyngeal and rectal temperature, arterial pressure in both radial arteries, perfusion rate and perfusion pressure during both of CPB and unilateral SACP, lowest hemoglobin concentration (g/L) and hematocrit (%), acid-base indices, intraoperative red blood cell transfusion (units), highest dose/agent used for intraoperative inotrope or vasopressor support. Also during the surgery will be performed NIRS and BIS-monitoring.

Postoperative data will include valuation of following indicators: mortality (hospital mortality and death from any cause); neurological injury (TIA, stroke, delirium), MRI and CT-scan only in event of postoperative stroke; acute kidney injury (creatinine level prior and 1, 2, 4 postoperative day (POD), urine output-up to 24-48 h, renal replacement therapy (dialysis); time of mechanical ventilation; re-exploration for bleeding, tamponade or other reasons; postoperative transfusion (packed red blood cells, platelets, fresh frozen platelets, cryoprecipitate); postoperative myocardial infarction (electrocardiogram and troponins); inotropic support during 24-48 h (agent and dose (VIS)); length of stay (intensive care unit and total hospital days).

Before surgery and on 12-16 POD, patients will undergo neurocognitive screening by trained personnel. Neurocognitive tests will include: MOCA examinations, Schulte Table and The Bourdon Test.

In addition, indicators of specific markers of brain damage will be evaluated. Indicators such as neuron-specific enolase (NSE), glial fibrillary acidic protein (GFAP), brain-derived neurotrophic factor (BDNF) will be evaluated before surgery and on first POD. Also will be evaluated indicators of the hemostatic system: thrombin-antithrombin (TAT) complexes, prothrombin fragments 1+2, glu-plasminogen, tissue plasminogen activator (t-PA), endothelin 1-21 and thromboelastography (TEG) in following points - before surgery, lowest temperature during arrest time, after inactivation of heparin and 4 h after surgery.

Follow-up information will be collected using direct or phone contact with patients, relatives, or physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ascending aortic aneurysm
* Elective aortic hemiarch replacement
* Able to provide written informed consent

Exclusion Criteria:

* Surgery for acute aortic dissection or emergent operations
* Patients with known/documented coagulopathy
* Oncological disease (high degrees)
* Severe chronic heart failure
* Refusal of surgical treatment
* Patients in renal failure or currently being treated with renal replacement therapy (RRT) or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
* Severe carotid disease, defined as: any patient with previously documented carotid stenosis of > 70%, without neurological deficits; or carotid stenosis > 50% with neurological deficits; or previous carotid endarterectomy or stenting
* Pre-existing severe neurological impairment or inability to accurately assess neurocognitive function as determined by the operating surgeon

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Operative mortality | During the first 30 days after the procedure
  Operative mortality (%) as assessed by data linkage to medical records Comparison of mild (30-32°C) vs moderate (26-28°C) hypothermia in aortic hemiarch surgery with respect to the incidence of death
Composite of neurologic injury | During the first 30 days after the procedure
  Percentage of patients with neurological complications is assessed. Single assessment by CT or MRI. More often if necessary. Comparison of mild (30-32°C) vs moderate (26-28°C) hypothermia in aortic hemiarch surgery with respect to incidence of neurologic injury, including transient ischemic attack (TIA), permanent neurological dysfunction (PND) or stroke and delirium
Incidence of Acute Kidney Injury (AKI) | During the first 30 days after the procedure
  The incidence of acute kidney injury (AKI) (%), defined as Stage 1 or greater using the KDIGO criteria. Using the KDIGO criteria, Stage 1 AKI is defined as an increase in serum creatinine of 1.5-1.9x the baseline or an increase >= 27umol/L with urine output <0.5 mL/kg/hour for 6-12 hours.

SECONDARY OUTCOMES:
Respiratory failure | During the first 30 days after the procedure
  Percentage of patients with respiratory failure. Artificial ventilation for more than 48 hours requiring tracheostomy during ICU stay of the patient as assessed by data linkage to medical records
Perioperative Myocardial Infarction | During the first 30 days after the procedure (assessed by daily serum assay and ECG in the ICU and every 5 days after discharge from ICU. )
  Incidence of the myocardial infarction (%) is assessed by complex evaluation based on the ECG and echocardiographic changes as well as increase of the troponin level using serum assay
Rates of re-exploration for bleeding | During the first 3 days after the procedure
  Percentage of patients requiring re-exploration for bleeding. Comparison of mild (30-32°C) vs moderate (26-28°C) hypothermia in aortic hemiarch surgery with respect to the rates of mediastinal re-exploration (re-operation) for bleeding.
Volume of perioperative blood transfusion | During the first 3 days after the procedure
  Defined as the volume (mL) of all intraoperative and postoperative blood transfusions
The duration of a patient's stay in the intensive care unit and on the hospital ward | Up to 90 days after surgery
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the duration of a patient's stay in the intensive care unit and on the hospital ward.
Duration of cardiopulmonary bypass | During the index procedure
  Differences in the duration of cardiopulmonary bypass used in patients who receive mild or moderate hypothermic circulatory arrest during aortic hemiarch surgery are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry S Panfilov, PhD, Principal Investigator — Tomsk National Research Medical Center of the Russian Academy of Sciences
Locations (1):
- Tomsk NRMC, Tomsk, Russia